CLINICAL TRIAL: NCT03354221
Title: A Pilot Study Assessing the Efficacy of Short Duration Six Food Elimination Diet in Eosinophilic Esophagitis (EoE)
Brief Title: Short Duration 6Fed Sponge For EoE Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in literature to suggest at least 6 weeks of initial elimination is necessary to see decrease in eosinophil count.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Karthik Ravi, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-002185
Record Dates: First submitted 2017-09-25; First posted 2017-11-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Eosinophilic Esophagitis
Keywords: EoE
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cytosponge, Diet, EEsAI Pro, Likert Scoring Scale (Experimental): Patients going through the six food elimination diet (clinically) for EoE will be asked to participate. During the initial 6 week elimination period, participants will return at 2, 4 and 6 weeks to swallow the cytosponge. The cytosponge is a 10 minute procedure done in the office. This will be sent for histology, <15 phf would be considered a responder. Results of the histology will help the investigator to direct the future of the 6 food elimination diet to determine if a period of 6 weeks of initial elimination is necessary. The EEsAI Pro questionnaire measures symptomatic response to the elimination of the foods. The Likert Scoring Scale measures patient experience of the cytosponge and the upper endoscopy.
  Interventions: Device: Cytosponge; Other: Diet; Other: EEsAI Pro; Other: Likert Scoring Scale

INTERVENTIONS:
Device: Cytosponge — Patients undergoing the six food elimination diet will be monitored during the initial elimination period at 2, 4 and 6 weeks with swallowing the cytosponge. This is a ten minute procedure in the office. The cytosponge will be sent to the lab for histology reading of the eosinophilic count.
  Other Names: sponge
Other: Diet — During the initial 6 week elimination period, participants will eliminate the 6 most common food allergens from their diet (fish, nuts, eggs, soy, wheat, dairy). Participants will return for the cytosponge during this time at 2, 4 and 6 weeks of elimination.
  Other Names: SFED, 6FED
Other: EEsAI Pro — This is a short questionnaire to assess the participants swallowing. This will be completed at baseline and during each cytosponge visit during the initial elimination period (2, 4, 6 weeks).
  Other Names: Eosinophilic Esophagitis Activity Index Pro questionnaire
Other: Likert Scoring Scale — This is a short questionnaire for patients to compare their experiences swallowing the cytosponge versus completing an upper endoscopy. The scale is rated from "worst experience" to "best experience."
  Other Names: Likert score

SUMMARY:
This research is being done to see if the investigators can use the cytosponge or esophacap (depending on availability) to determine if shorter duration SFED (two weeks versus six weeks) would have equal results.

DETAILED DESCRIPTION:
Dietary therapy has been shown to be successful in the treatment of adult and pediatric patients with eosinophilic esophagitis (EoE). Dietary studies were initially reported in children, but the results appear to be similar in adult patients. Elemental diets are successful in 70-95% of patients but are poorly tolerated.

The six food elimination diet (SFED) involves the elimination of the six most common food allergens (i.e. milk, wheat, soy, eggs, nuts, and fish) for six weeks and has become the mainstay of dietary therapy in EoE. A six week SFED has demonstrated excellent efficacy and durability in both pediatric and adult EoE. However, compliance with the SFED for a total of six weeks can be challenging for patients.

Previous studies have found the esophageal sponge to be an accurate technique of accessing esophageal eosinophilia in EoE . The sponge is swallowed as a 12 mm capsule on a string. The capsule rapidly dissolves upon entering the stomach and the sponge then expands and can be pulled out the mouth five minutes after ingestion. In previous studies, the procedure was very well tolerated and all patients preferred the sponge to endoscopy. Therefore the sponge is a well tolerated, inexpensive, very low risk procedure that would be an ideal option to replace EGD esophageal sampling in the evaluation of dietary treatment of EoE.

Although initially described as a six week trial, it is possible that a shorter duration food elimination diet of 2 or 4 weeks would have equal efficacy. This would have important implications for patients as it would make the diet more tolerable.

ELIGIBILITY:
Inclusion criteria:

* Adults ages 18-70 years of age
* Diagnosis of EoE, i.e. symptoms of esophageal dysfunction with histologic finding of 15 or more eosinophils per high power field on esophageal biopsy despite 8 weeks of high dose proton pump inhibitor therapy.
* Scheduled to initiate a clinical SFED for treatment of EoE

Exclusion criteria:

* Clinical evidence of infectious process potentially contributing to dysphagia (e.g. candidiasis, CMV, herpes)
* Other cause of dysphagia identified at endoscopy (e.g. reflux esophagitis, stricture, web, ring, achalasia, esophageal neoplasm)
* Esophageal minimal diameter < 13 mm on structured barium esophagram
* Inability to read due to: Blindness, cognitive dysfunction, or English language illiteracy
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Cytosponge pathology: number of Eosinophils directing dietary therapy | 2 years
  Patients will swallow the cytosponge at 2 weeks, 4 weeks and 6 weeks into the initial period of the 6 food elimination diet. Eosinophils <15 phf will be considered histologic remission to dietary therapy. This response will be compared to the 6 week visit sponge eosinophilic histology.

SECONDARY OUTCOMES:
Eosinophilic Esophgitis Activity Index Pro (EEsAI Pro) | 2 years
  The EEsAI Pro uses the VDQ is visual dysphagia question AMS is avoidance, modification, slow eating question. Thes two along with questions on frequency of, duration of, pain associated with dysphagia make up the PRO (patient reported outcomes). The PRO is a number (0-100) calculated from the answer to the questions. A PRO<20 defines asymptomatic EoE.
The tolerability of esophageal sponge compared to upper endoscopy with biopsy. | 6 weeks
  Patients return at the end of the 6 weeks initial elimination of the diet will complete the modified Likert scoring scale. This scale rates participant experience of the cytosponge versus the upper endoscopy. This is a short questionnaire for patients to compare their experiences swallowing the cytosponge versus completing an upper endoscopy. The scale is rated from "worst experience" to "best experience."

CONTACTS AND LOCATIONS:
Overall Officials: Karthik Ravi, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Background] Aceves SS, Ackerman SJ. Relationships between eosinophilic inflammation, tissue remodeling, and fibrosis in eosinophilic esophagitis. Immunol Allergy Clin North Am. 2009 Feb;29(1):197-211, xiii-xiv. doi: 10.1016/j.iac.2008.10.003. PMID 19141355
- [Background] Kelly KJ, Lazenby AJ, Rowe PC, Yardley JH, Perman JA, Sampson HA. Eosinophilic esophagitis attributed to gastroesophageal reflux: improvement with an amino acid-based formula. Gastroenterology. 1995 Nov;109(5):1503-12. doi: 10.1016/0016-5085(95)90637-1. PMID 7557132
- [Background] Liacouras CA, Spergel JM, Ruchelli E, Verma R, Mascarenhas M, Semeao E, Flick J, Kelly J, Brown-Whitehorn T, Mamula P, Markowitz JE. Eosinophilic esophagitis: a 10-year experience in 381 children. Clin Gastroenterol Hepatol. 2005 Dec;3(12):1198-206. doi: 10.1016/s1542-3565(05)00885-2. PMID 16361045
- [Background] Peterson KA, Byrne KR, Vinson LA, Ying J, Boynton KK, Fang JC, Gleich GJ, Adler DG, Clayton F. Elemental diet induces histologic response in adult eosinophilic esophagitis. Am J Gastroenterol. 2013 May;108(5):759-66. doi: 10.1038/ajg.2012.468. Epub 2013 Feb 5. PMID 23381017
- [Background] Gonsalves N, Yang GY, Doerfler B, Ritz S, Ditto AM, Hirano I. Elimination diet effectively treats eosinophilic esophagitis in adults; food reintroduction identifies causative factors. Gastroenterology. 2012 Jun;142(7):1451-9.e1; quiz e14-5. doi: 10.1053/j.gastro.2012.03.001. Epub 2012 Mar 3. PMID 22391333
- [Background] Lucendo AJ, Arias A, Gonzalez-Cervera J, Yague-Compadre JL, Guagnozzi D, Angueira T, Jimenez-Contreras S, Gonzalez-Castillo S, Rodriguez-Domingez B, De Rezende LC, Tenias JM. Empiric 6-food elimination diet induced and maintained prolonged remission in patients with adult eosinophilic esophagitis: a prospective study on the food cause of the disease. J Allergy Clin Immunol. 2013 Mar;131(3):797-804. doi: 10.1016/j.jaci.2012.12.664. Epub 2013 Jan 31. PMID 23375693
- [Background] Kagalwalla AF, Shah A, Li BU, Sentongo TA, Ritz S, Manuel-Rubio M, Jacques K, Wang D, Melin-Aldana H, Nelson SP. Identification of specific foods responsible for inflammation in children with eosinophilic esophagitis successfully treated with empiric elimination diet. J Pediatr Gastroenterol Nutr. 2011 Aug;53(2):145-9. doi: 10.1097/MPG.0b013e31821cf503. PMID 21788754
- [Background] Arias A, Gonzalez-Cervera J, Tenias JM, Lucendo AJ. Efficacy of dietary interventions for inducing histologic remission in patients with eosinophilic esophagitis: a systematic review and meta-analysis. Gastroenterology. 2014 Jun;146(7):1639-48. doi: 10.1053/j.gastro.2014.02.006. Epub 2014 Feb 15. PMID 24534634
- [Background] Molina-Infante J, Arias A, Barrio J, Rodriguez-Sanchez J, Sanchez-Cazalilla M, Lucendo AJ. Four-food group elimination diet for adult eosinophilic esophagitis: A prospective multicenter study. J Allergy Clin Immunol. 2014 Nov;134(5):1093-9.e1. doi: 10.1016/j.jaci.2014.07.023. Epub 2014 Aug 28. PMID 25174868
- [Background] Katzka DA, Geno DM, Ravi A, Smyrk TC, Lao-Sirieix P, Miremadi A, Debiram I, O'Donovan M, Kita H, Kephart GM, Kryzer LA, Camilleri M, Alexander JA, Fitzgerald RC. Accuracy, safety, and tolerability of tissue collection by Cytosponge vs endoscopy for evaluation of eosinophilic esophagitis. Clin Gastroenterol Hepatol. 2015 Jan;13(1):77-83.e2. doi: 10.1016/j.cgh.2014.06.026. Epub 2014 Jul 3. PMID 24997328
- [Background] Dellon ES, Gonsalves N, Hirano I, Furuta GT, Liacouras CA, Katzka DA; American College of Gastroenterology. ACG clinical guideline: Evidenced based approach to the diagnosis and management of esophageal eosinophilia and eosinophilic esophagitis (EoE). Am J Gastroenterol. 2013 May;108(5):679-92; quiz 693. doi: 10.1038/ajg.2013.71. Epub 2013 Apr 9. PMID 23567357
- [Background] Schoepfer AM, Straumann A, Panczak R, Coslovsky M, Kuehni CE, Maurer E, Haas NA, Romero Y, Hirano I, Alexander JA, Gonsalves N, Furuta GT, Dellon ES, Leung J, Collins MH, Bussmann C, Netzer P, Gupta SK, Aceves SS, Chehade M, Moawad FJ, Enders FT, Yost KJ, Taft TH, Kern E, Zwahlen M, Safroneeva E; International Eosinophilic Esophagitis Activity Index Study Group. Development and validation of a symptom-based activity index for adults with eosinophilic esophagitis. Gastroenterology. 2014 Dec;147(6):1255-66.e21. doi: 10.1053/j.gastro.2014.08.028. Epub 2014 Aug 23. PMID 25160980
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials